CLINICAL TRIAL: NCT02998450
Title: A Phase 1a Study of IMR-687 in Healthy Adult Volunteers
Brief Title: A Study of IMR-687 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cardurion Pharmaceuticals, Inc. (Industry)
Collaborators: Quintiles, Inc. (Industry); Imara, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMR-SCD-101
Record Dates: First submitted 2016-12-06; First posted 2016-12-20 (Estimated); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Sickle Cell Disease; Sickle-Cell; Hb-SC; Sickle Beta 0 Thalassemia
Keywords: Sickle Cell Disease; Sickle Beta 0 Thalassemia
MeSH Terms: conditions — Anemia, Sickle Cell; Hemoglobin SC Disease | interventions — microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1 (Experimental): 4 Subjects will receive a single low dose of IMR-687, administered orally following an overnight fast.
  2 Subjects will receive a single dose of Placebo, administered orally following an overnight fast.
  Interventions: Drug: IMR-687; Drug: Placebo Oral Capsule
- Cohort 2 (Experimental): 4 Subjects will receive a single low-mid dose of IMR-687, administered orally following an overnight fast.
  2 Subjects will receive a single dose of Placebo, administered orally following an overnight fast.
  Interventions: Drug: IMR-687; Drug: Placebo Oral Capsule
- Cohort 3 (Experimental): 4 Subjects will receive a single mid-low dose of IMR-687, administered orally following an overnight fast.
  2 Subjects will receive a single dose of Placebo, administered orally following an overnight fast.
  Interventions: Drug: IMR-687; Drug: Placebo Oral Capsule
- Cohort 4 (Experimental): 4 Subjects will receive a single mid dose of IMR-687, administered orally following an overnight fast.
  2 Subjects will receive a single dose of Placebo, administered orally following an overnight fast.
  Interventions: Drug: IMR-687; Drug: Placebo Oral Capsule
- Cohort 5 (Experimental): 4 Subjects will receive a single mid-high dose of IMR-687, administered orally following an overnight fast.
  2 Subjects will receive a single dose of Placebo, administered orally following an overnight fast.
  Interventions: Drug: IMR-687; Drug: Placebo Oral Capsule
- Cohort 6 (Experimental): 4 Subjects will receive a single high dose of IMR-687, administered orally following an overnight fast.
  2 Subjects will receive a single dose of Placebo, administered orally following an overnight fast.
  Interventions: Drug: IMR-687; Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: IMR-687 — 1 of 6 possible single doses administered orally following overnight fast
Drug: Placebo Oral Capsule — Placebo oral capsule with 50 mg microcrystalline cellulose in capsules identical to those used for the active pharmaceutical ingredient.
  Other Names: Microcrystalline cellulose

SUMMARY:
The purpose of this Phase 1a, first in human, randomized, double-blind, placebo-controlled study is to evaluate the safety, tolerability, PK and PD profile of the orally administered IMR-687 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Be healthy as judged by the Investigator on the basis of pre-study tests performed at Screening, with healthy body mass index (BMI), healthy body weight, and laboratory results within normal laboratory reference range or determined not to be clinically significant by the Investigator; and be free from drugs of abuse.

Exclusion Criteria:

* Females who are pregnant, trying to become pregnant, or breastfeeding; and males with female partners who are trying to conceive.
* Asthmatics or other individuals who use or may use albuterol rescue inhalers or nebulizers.
* A significant history of cardiovascular disease.
* On ECG, a QTcF >450 ms or the presence of clinically significant abnormalities as determined by the Investigator.
* Elevated blood pressure.
* Use within 30 days prior to Day 1 of any inhibitors or substrates of targets of IMR-687.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2016-10-18 (Actual); Primary Completion 2017-07-08 (Actual); Study Completion 2017-07-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment emergent adverse events and serious adverse events | 5 Days
Number of participants with clinically significant changes from baseline in vital signs | Baseline to Day 5
  Vital signs include blood pressure, heart rate, pulse rate, and oral temperature
Number of participants with clinically significant changes from baseline in physical examination | Baseline to Day 5
Number of participants with clinically significant changes from baseline in hematology, chemistry, coagulation and urinalysis laboratory values | Baseline to Day 5
Number of participants with clinically significant changes from baseline in 12-lead ECG parameters | Baseline to Day 2
Use of concomitant medications and therapies, medication type and frequency | 5 Days

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of IMR-687 | Day 1 prior to administration of drug and 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 24 hours post dose
  Maximum Observed Plasma Concentration (Cmax) of IMR-687
Pharmacokinetics (PK) of IMR-687 | Day 1 prior to administration of drug and 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 24 hours post dose
  Area under the curve (AUC) ( 0 to 24 h) of IMR-687
Pharmacokinetics (PK) of IMR-687 | Day 1 prior to administration of drug and 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 24 hours post dose
  AUC from time 0 to the last measurable time point (AUClast) of IMR-687
Pharmacokinetics (PK) of IMR-687 | Day 1 prior to administration of drug and 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 24 hours post dose
  AUC extrapolated to infinity (AUC0 ∞) of IMR-687
Pharmacokinetics (PK) of IMR-687 | Day 1 prior to administration of drug and 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 24 hours post dose
  Time to maximum concentration (tmax) of IMR-687
Pharmacokinetics (PK) of IMR-687 | Day 1 prior to administration of drug and 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 24 hours post dose
  Apparent terminal half-life (t½) of IMR-687
The change from baseline in QTcF interval. | 2 Days

CONTACTS AND LOCATIONS:
Overall Officials: Regulatory Operations, Study Director — Cardurion Pharmaceuticals
Locations (1):
- Quintiles, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No